CLINICAL TRIAL: NCT01483690
Title: A Pilot Study of Decitabine and Vorinostat With Chemotherapy for Relapsed ALL
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Toxicity
Sponsor: Therapeutic Advances in Childhood Leukemia Consortium (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T2009-003
Record Dates: First submitted 2011-11-29; First posted 2011-12-01 (Estimated); Results first posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Acute Lymphoblastic Leukemia; Precursor B-Cell Lymphoblastic Leukemia; Precursor T-Cell Lymphoblastic Leukemia
Keywords: Relapse; Lymphoblastic; Leukemia; Decitabine; Vorinostat; Refractory; Acute; Childhood; Pediatric; ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor B-Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Recurrence; Leukemia | interventions — Decitabine; Vorinostat; Vincristine; Dexamethasone; Calcium Dobesilate; dexamethasone acetate; dexamethasone 21-phosphate; Mitoxantrone; pegaspargase; Methotrexate; merphos

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Initial Dose Level (Experimental): Decitabine 15 mg/m2/day given IV over 1 hour on days 1 through 7 and days 15 through 21.
  Vorinostat: 180 mg/m2/day (Max dose=400 mg daily) given orally on days 3 through 10 and days 17 through 24
  Interventions: Drug: Decitabine; Drug: Vorinostat; Drug: Vincristine; Drug: Dexamethasone; Drug: Mitoxantrone; Drug: Pegaspargase; Drug: Methotrexate
- Modified Dose Level (Experimental): Decitabine 10 mg/m2/day given IV over 1 hour on days 1 through 5 and days 15 through 19.
  Vorinostat: 180 mg/m2/day (Max dose=400 mg daily) given orally on days 2 through 7 and days 16 through 21
  Interventions: Drug: Decitabine; Drug: Vorinostat; Drug: Vincristine; Drug: Dexamethasone; Drug: Mitoxantrone; Drug: Pegaspargase; Drug: Methotrexate

INTERVENTIONS:
Drug: Decitabine — 10 mg/m2/day given IV over 1 hour on days 1 through 5 and days 15 through 19.
  Other Names: Dacogen
Drug: Vorinostat — 180 mg/m2/day (Max dose=400mg daily) given orally on days 2 through 7 and days 16 through 21.
  Other Names: Zolinza; suberoylanilide hydroxamic acid (SAHA)
Drug: Vincristine — 1.5 mg/m2/day (Max dose 2 mg) given IV push on days 10, 17, 24 and 31.
  Other Names: Oncovin; Vincasar PFS; Vincrex; vincristine sulfate; VCR
Drug: Dexamethasone — 20 mg/m2/day divided BID given orally on days 8 through 12 and 22 through 26.
  Other Names: Decadron; Dexamethasone Intensol; dexamethasone acetate; dexamethasone sodium phosphate
Drug: Mitoxantrone — 10 mg/m2/day given on days 8 and 9 as a short IV infusion over 5-15 minutes; do not infuse over less than 3 minutes
  Other Names: Novantrone; DHAD; DHAQ
Drug: Pegaspargase — 2500 international units/m2/day IM or IV on days 10 and 24.
  Other Names: Oncospar; PEG-L-asparaginase
Drug: Methotrexate — Given intrathecally to all patients the dose defined by age below.
  * 8 mg for patients age 1-1.99
  * 10 mg for patients age 2-2.99
  * 12 mg for patients 3-8.99 years of age
  * 15 mg for patients >9 years of age
  CNS 1 or 2 patients get doses on day 8, 22 and 35 and CNS 3 patients should get doses on day 8, 15, 22, 29 and 35
  Other Names: Folex; Mexate; MTX; Methotrex

SUMMARY:
This is a pilot study using decitabine and vorinostat before and during chemotherapy with vincristine, dexamethasone, mitoxantrone, and peg-asparaginase in pediatric patients with acute lymphoblastic leukemia (ALL).

DETAILED DESCRIPTION:
Decitabine is a demethylating agent and vorinostat is a HDAC inhibitor. The use of demethylating agents and HDAC inhibitors in combination have been previously shown to have synergistic effects in altering neoplastic pathways of cancer cells and be well tolerated in human clinical studies. With the ability of decitabine and vorinostat to alter the abnormal cellular pathways of leukemic blasts and essentially turn off anti-apoptotic proteins, the leukemia cells have become primed for cytotoxic cell kill via chemotherapeutic agents. This study will ask the question as to whether or not the combination of decitabine and vorinostat followed by chemotherapy is feasible and whether it can positively impact outcome in patients with relapsed or refractory acute lymphoblastic leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥1 and ≤ 21 years of age when originally diagnosed with ALL.

Diagnosis

* Patients must have a diagnosis of acute lymphoblastic leukemia (ALL) with ≥ 25% blasts in the bone marrow (M3), with or without extramedullary disease.
* Patients may have CNS 1, 2 or 3 disease.
* Karnofsky > 50% for patients > 16 years of age and Lansky > 50% for patients ≤ 16 years of age.
* Prior Therapy
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.
* Patients must have had 2 or more prior therapeutic attempts defined as:
* Relapse after going into remission from re-induction for the first or subsequent relapse (ie: 2nd , 3rd, 4th…relapse), OR
* Refractory disease after first or greater relapse and a re-induction attempt, OR
* Failing to go into remission from original diagnosis after 2 previous induction attempts.
* Hematopoietic Stem Cell Transplant: Patients who have experienced their relapse after a HSCT are eligible, provided they have no evidence of Graft-versus-Host Disease (GVHD) and are at least 60 days post-transplant at the time of enrollment.
* Prior anthracycline exposure: Patients must have less than 400 mg/m2 lifetime exposure of anthracycline chemotherapy. (See Appendix II for calculation worksheet)
* Hematopoietic grow factors: It must have been at least 7 days since the completion of therapy with GCSF or other growth factors at the time of enrollment. It must have been at least 14 days since the completion of therapy with pegfilgrastim (Neulasta®).
* Biologic (anti-neoplastic) therapy: It must be at least 7 days after last does of biologic agent. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair
* Monoclonal antibodies: At least 3 half-lives of the antibody must have elapsed after the last dose of monoclonal antibody. (ie. Rituximab=66 days, Epratuzumab=69 days)
* Immunotherapy: At least 42 days after the completion of any type of immunotherapy, e.g. tumor vaccines.

Renal and Hepatic Function

* Patient's serum creatinine must be ≤ 1.5 x institutional upper limit of normal (ULN) according to age. If the serum creatinine is greater than 1.5 times normal, the patient must have a calculated creatinine clearance or radioisotope GRF ≥ 70mL/min/1.73m2.
* Patient's ALT and AST must be < 5 x institutional upper limit of norm ULN. The hepatic requirements are waived for patients with known or suspected liver involvement who would otherwise be eligible after consultation with the Study Chair or Vice Chair.
* Patient's total bilirubin must be ≤ 1.5 x ULN. The hepatic requirements are waived for patients with known or suspected liver involvement who would otherwise be eligible.

Cardiac Function:

* Patient must have a shortening fraction ≥ 27% by Echo or an ejection fraction ≥ 50% by MUGA.

Reproductive Function

* Female patients of childbearing potential must have a negative urine or serum pregnancy test confirmed prior to enrollment.
* Female patients with infants must agree not to breastfeed their infants while on this study.
* Male and female patients of child-bearing potential must agree to use an effective method of contraception approved by the investigator during the study.

Exclusion Criteria:

* Patients will be excluded if they are receiving Valproic Acid (VPA) therapy.
* Patients will be excluded if they have a known allergy to any of the drugs used in the study.
* Patients will be excluded if they have a systemic fungal, bacterial, viral or other infection that is exhibiting ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics or other treatment.
* Patients will be excluded if there is a plan to administer non-protocol chemotherapy, radiation therapy, or immunotherapy during the study period.
* Patients will be excluded if they have significant concurrent disease, illness, psychiatric disorder or social issue that would compromise patient safety or compliance with the protocol treatment or procedures, interfere with consent, study participation, follow up, or interpretation of study results.
* Patients will be excluded if they have had any positive fungal culture in the last 30 days prior to enrollment.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2011-12; Primary Completion 2015-07-31 (Actual); Study Completion 2015-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Burke, MD, Study Chair — Medical College of Wisconsin
Locations (28):
- United States (25):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - CHOC, Orange, California
  - UCSF School of Medicine, San Francisco, California
  - The Children's Hospital, University of Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Miami Cancer Center, Miami, Florida
  - Children's Healthcare of Atlanta, Emory University, Atlanta, Georgia
  - Lurie Children's Hospital, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Dana Farber, Boston, Massachusetts
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Childrens Hospital & Clinics of Minnesota, Minneapolis, Minnesota
  - University of Minnesota Children's Hospital, Minneapolis, Minnesota
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - New York University Medical Center, New York, New York
  - Children's Hospital New York-Presbyterian, New York, New York
  - Levine Children's Hospital at Carolinas Medical Center, Charlotte, North Carolina
  - Nationwide Childrens Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude, Memphis, Tennessee
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - University of Texas at Southwestern, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Australia (3):
  - Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Children's Hospital, Brisbane, Queensland
  - Sydney Children's Hospital, Sydney

REFERENCES:
- [Derived] Burke MJ, Kostadinov R, Sposto R, Gore L, Kelley SM, Rabik C, Trepel JB, Lee MJ, Yuno A, Lee S, Bhojwani D, Jeha S, Chang BH, Sulis ML, Hermiston ML, Gaynon P, Huynh V, Verma A, Gardner R, Heym KM, Dennis RM, Ziegler DS, Laetsch TW, Oesterheld JE, Dubois SG, Pollard JA, Glade-Bender J, Cooper TM, Kaplan JA, Farooqi MS, Yoo B, Guest E, Wayne AS, Brown PA. Decitabine and Vorinostat with Chemotherapy in Relapsed Pediatric Acute Lymphoblastic Leukemia: A TACL Pilot Study. Clin Cancer Res. 2020 May 15;26(10):2297-2307. doi: 10.1158/1078-0432.CCR-19-1251. Epub 2020 Jan 22. PMID 31969338
- [Derived] Raetz EA, Bhatla T. Where do we stand in the treatment of relapsed acute lymphoblastic leukemia? Hematology Am Soc Hematol Educ Program. 2012;2012:129-36. doi: 10.1182/asheducation-2012.1.129. PMID 23233571
- See also: Therapeutic Advances in Childhood Leukemia & Lymphoma Consortium web site. — http://www.tacl.us

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a pilot study where 16 patients are anticipated to be enrolled. Anticipated enrollment will take 2.5 years.
Period: Overall Study
Arm/Group | Initial Dose Level | Modified Dose Level
Started | 5 | 18
Completed | 3 | 13
Not Completed | 2 | 5
Not completed — Adverse Event | 1 | 2
Not completed — clinical deterioration | 1 | 0
Not completed — Physician Decision | 0 | 2
Not completed — exclusionary procedure | 0 | 1

BASELINE CHARACTERISTICS:
Population: Total number of participants enrolled into the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Initial Dose Level | Modified Dose Level | Total
Number analyzed (Participants) | 5 | 18 | 23
Age, Continuous [Median (Full Range); unit: years] | 12.5 [4.9 to 14.5] | 12.0 [1.6 to 21.4] | 12.0 [1.6 to 21.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 3 | 14 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 9 | 12
  Not Hispanic or Latino | 2 | 9 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 5 | 10 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 5 | 5
CNS Status [Count of Participants; unit: Participants] — Central nervous system (CNS) disease is divided into the following:
  CNS 1 - no evidence of leukemia cerebral spinal fluid (CSF)(best outcome) CNS 2 - <5 WBC in CSF with blasts present CNS 3 - > or = 5 WBC in CSF with blasts present (worse outcome).
  Participants
    CNS 1 | 4 | 14 | 18
    CNS 2 | 1 | 2 | 3
    CNS 3 | 0 | 2 | 2
Prior hematopoietic cell transplantation (HCT) [Count of Participants; unit: Participants]
  Yes had prior HCT | 3 | 8 | 11
  No did not have prior HCT | 2 | 10 | 12
Relapse # at enrollment [Count of Participants; unit: Participants]
  2nd Relapse | 2 | 13 | 15
  3rd Relapse | 1 | 1 | 2
  Refractory | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Dose Limiting Toxicity (DLT).
Description: To evaluate the side effects of giving decitabine and vorinostat before and during chemotherapy using the standard drugs vincristine, dexamethasone, PEG-asparaginase and mitoxantrone.
Time Frame: 6 weeks
Population: Participants who entered the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Initial Dose Level | Modified Dose Level
Number analyzed (Participants) | 5 | 18
Participants
  # of patients with DLT | 2 | 1
  # of patients without DLT | 2 | 12
  # of patients not evaluable | 1 | 5

2. Secondary Outcome: Disease Response Rate After Treatment.
Description: Bone marrow evaluation was performed on Day 35 of study to evaluate treatment response. CR defined as attaining M1 marrow (<5% blasts) with no evidence of circulating blasts or extramedullary disease in addition to recovery of peripheral blood counts (ANC >750/uL and platelet count >75,000/uL). CRp was defined as attaining an M1 marrow with no evidence of circulating blasts or extramedullary disease in addition to recovery of ANC but insufficient recovery of platelets. CRi was attaining M1 marrow with no evidence of circulating blasts or extramedullary disease but insufficient recovery of ANC with or without sufficient recovery of platelets. PR was defined as no evidence of circulating blasts and achievement of M2 marrow (5-25% blasts) without new sites of disease and with recovery of ANC. SD is for patients who did not meet the criteria for PR, CR, CRp, or CRi. PD is an increase of at least 25% in the absolute number of leukemia cells or development of new sites.
Time Frame: 6 weeks
Population: Patients who entered the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Initial Dose Level | Modified Dose Level
Number analyzed (Participants) | 5 | 18
Participants
  complete response (CR) | 0 | 1
  complete response without platelet recovery (CRp) | 1 | 3
  complete remission with incomplete recovery (CRi) | 1 | 3
  stable disease (SD) | 1 | 4
  patient not evaluable for response | 2 | 7

ADVERSE EVENTS:
Time Frame: Adverse events and suspected adverse reactions will be collected and reported on the electronic case report forms beginning with the first dose of decitabine and vorinostat until 30 days following last dose of decitabine and vorinostat.
Description: The definition of adverse event and/or serious adverse event used to collect adverse event information is the same from clinicaltrials.gov definitions.
Arm/Group | Initial Dose Level | Modified Dose Level
All-Cause Mortality (participants affected / at risk) | 5/5 | 13/18
Serious Adverse Events (participants affected / at risk) | 5/5 | 18/18
Other Adverse Events (participants affected / at risk) | 5/5 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Initial Dose Level (N=5) | Modified Dose Level (N=18)
Anemia (Metabolism and nutrition disorders) | 1 | 11
Acidosis (Metabolism and nutrition disorders) | 0 | 2
Acute kidney injury (Endocrine disorders) | 0 | 2
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Agitation (Musculoskeletal and connective tissue disorders) | 0 | 1
Alanine aminotransferase increase (Metabolism and nutrition disorders) | 0 | 2
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 0 | 3
Ano-rectal infection (Infections and infestations) | 0 | 1
Blood bilirubin increased (Metabolism and nutrition disorders) | 1 | 2
Encephalopathy (Nervous system disorders) | 0 | 1
GGT increased (Metabolism and nutrition disorders) | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatermia (Metabolism and nutrition disorders) | 1 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 2 | 9
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 2
Hypotension (Cardiac disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Left ventricular systolic dysfunction (Cardiac disorders) | 1 | 1
Lipase increased (Metabolism and nutrition disorders) | 1 | 2
Lung infection (Infections and infestations) | 0 | 1
Lymphocyte count decreased (Metabolism and nutrition disorders) | 2 | 2
Lymphocyte count increased (Metabolism and nutrition disorders) | 0 | 1
nervous system disorder - other (Nervous system disorders) | 0 | 1
neutrophil count decrease (Blood and lymphatic system disorders) | 2 | 5
Altered mental status (Nervous system disorders) | 0 | 1
platelet count decreased (Blood and lymphatic system disorders) | 2 | 7
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 | 1
sepsis (Infections and infestations) | 2 | 4
serum amylase increased (Metabolism and nutrition disorders) | 0 | 1
sinus bradycardia (Cardiac disorders) | 0 | 2
soft tissue infection (Infections and infestations) | 0 | 1
white blood cell decreased (Blood and lymphatic system disorders) | 2 | 6
Bone marrow hypocellular (Blood and lymphatic system disorders) | 1 | 0
Capillary leak syndrome (Blood and lymphatic system disorders) | 1 | 0
Gastrointestinal disorder - Other (Gastrointestinal disorders) | 1 | 0
Right ventricular dysfunction (Cardiac disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Somnolence (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Initial Dose Level (N=5) | Modified Dose Level (N=18)
Abdominal pain (Gastrointestinal disorders) | 3 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 1 | 3
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 15
Anorexia (General disorders) | 2 | 4
Ascites (Gastrointestinal disorders) | 0 | 1
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 1 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Blood bilirubin increased (Blood and lymphatic system disorders) | 1 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Catheter related infection (Infections and infestations) | 1 | 3
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cholesterol high (Metabolism and nutrition disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Creatinine increased (Metabolism and nutrition disorders) | 0 | 2
Dehydration (General disorders) | 1 | 1
Delirium (General disorders) | 1 | 1
Depressed level of consciousness (General disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 2
Dizziness (General disorders) | 0 | 1
Dyspnea (General disorders) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 2
Epistaxis (General disorders) | 0 | 1
Febrile neutropenia (Infections and infestations) | 2 | 15
Fever (General disorders) | 1 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 2
Generalized muscle weakness (General disorders) | 1 | 2
Gamma-glutamyl transferase increased (Metabolism and nutrition disorders) | 1 | 0
Hepatobiliary disorders - Other (Gastrointestinal disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 3
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hypertension (Cardiac disorders) | 2 | 3
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 5
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 2 | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 6
Hypotension (Cardiac disorders) | 1 | 2
Hypoxia (General disorders) | 1 | 3
Ileus (Gastrointestinal disorders) | 0 | 1
Iron overload (Metabolism and nutrition disorders) | 0 | 1
Infective myositis (Infections and infestations) | 1 | 0
Investigations - Other (Investigations) | 1 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 1
Lethargy (General disorders) | 1 | 0
Lip infection (Infections and infestations) | 0 | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 1
Lung infection (Infections and infestations) | 1 | 4
Lymph gland infection (Infections and infestations) | 0 | 1
Lymphocyte count decreased (Metabolism and nutrition disorders) | 0 | 3
Lymphocyte count increased (Metabolism and nutrition disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Mucosal infection (Infections and infestations) | 1 | 2
Muscle weakness (General disorders) | 0 | 1
Nausea (General disorders) | 1 | 2
Pain in extremity (General disorders) | 0 | 2
Hyperammonemia (Metabolism and nutrition disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 3
Tumor lysis syndrome (Blood and lymphatic system disorders) | 1 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 1
Scrotal infection (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 2
Soft tissue infection (Infections and infestations) | 0 | 3
Spasticity (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Typhlitis (Infections and infestations) | 0 | 2
Weight loss (General disorders) | 0 | 2
White blood cell decreased (Blood and lymphatic system disorders) | 0 | 1
Coagulase negative staphylococus (Infections and infestations) | 1 | 0
Enterococcus Faecalis (Infections and infestations) | 2 | 0
Candida Kruseli (Infections and infestations) | 3 | 0
Klebsiella pneumonae (Infections and infestations) | 0 | 1
Candida parapsilosis (Infections and infestations) | 0 | 1
Pseudomonas aeruginosa (Infections and infestations) | 0 | 1
Necrotizing fascitis (Infections and infestations) | 0 | 1
Bipolaris spicifera (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days